CLINICAL TRIAL: NCT04261270
Title: A Randomized,Open,Controlled Small Sample Clinical Study to Evaluate the Efficacy and Safety of ASC09/Ritonavir Compound Tablets and Ritonavir for 2019-nCoV Pneumonia
Brief Title: A Randomized,Open,Controlled Clinical Study to Evaluate the Efficacy of ASC09F and Ritonavir for 2019-nCoV Pneumonia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASC09F-CTP-TJ-01
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: 2019-nCoV Pneumonia
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASC09F+Oseltamivir (Experimental)
  Interventions: Drug: ASC09F+Oseltamivir
- Ritonavir+Oseltamivir (Experimental)
  Interventions: Drug: Ritonavir+Oseltamivir
- Oseltamivir (Experimental)
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: ASC09F+Oseltamivir — ASC09F tablets:one tablet(400mg/tablet)twice a day for 14 days;Oseltamivir tablet:75mg,once a day
  Arms: ASC09F+Oseltamivir
Drug: Ritonavir+Oseltamivir — Ritonavir tablet:three tablets(100mg/tablet)twice a day for 14 days;Oseltamivir tablet:75mg,once a day
  Arms: Ritonavir+Oseltamivir
Drug: Oseltamivir — 75mg ,once a day
  Arms: Oseltamivir

SUMMARY:
Based on oseltamivir treatment, evaluate the efficacy and safety of ASC09/ritonavir compound tablets(ASC09F) or ritonavir tablets for 2019-nCoV infection patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18~55 years old, unlimited gender.
2. Laboratory (RT-PCR) confirmed infection with 2019-nCoV and accompanied with clinical manifestations.
3. Patients with newly diagnosed respiratory discomfort who have been hospitalized (The proper diagnosis time is less than 7 days).
4. Women who have no planned pregnancy in the next six months,and are willing to take effective measures to prevent contraception from the first dose of study drug to 30 days after the last dose.
5. Agree not to participate in other clinical studies within 30 days from the first dose of the study drug to the last dose.
6. Patients who voluntarily sign informed consent forms.

Exclusion Criteria:

1.2019-nCoV severe Pneumonia patients.

Meet the definition of severe pneumonia(Comply with any of the followings):

1. Respiratory distress ,RR≥30 bpm;
2. In a resting state:SPO2≤93%;
3. PaO2/ FiO2≤300mmHg.

   2.2019-nCoV critical and severe Pneumonia patients.Comply with any of the followings:Respiratory failure and need mechanical ventilation;Shock;Patients combined with other organ failure need ICU monitoring and treatment.

   3.Severe liver disease(such as:the ChildPugh score≥C;AST > 5 times the upper limit).

   4.Patients who are allergic to the ingredients of ASC09/ritonavir compound tablets.

   5.Patients with definite contraindications in ritonavir tablets.

   6.Female subjects were positive for the pregnancy test during the screening period.

   7.Researcher judges unsuitable for participation in this clinical trial(such as:during the study patients may be transferred to hospital for treatment;patients with multiple underlying diseases, etc)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of comprehensive adverse outcome | 14 days
  The definition of comprehensive adverse outcome is as follows:
  1. SPO2≤93% without oxygen inhalation;
  2. PaO2/FiO2≤300mmHg;
  3. RR≥30 bpm without oxygen inhalation.

SECONDARY OUTCOMES:
Time of clinical remission | 28 days
  The definition of clinical remission:
  1. Based on the symptoms of the disease (fever,cough,diarrhea,myalgia,dyspnea) has been relieved for 48 hours;
  2. There is no evidence of disease progression(New dyspnea, SpO2 decreased≥3%,RR≥30 bpm without oxygen inhalation).
Rate of no fever | 14 days
Rate of no cough | 14 days
Rate of no dyspnea | 14 days
Rate of no need for oxygen inhalation | 14 days
Rate of undetectable viral RNA | 14 days
Rate of mechanical ventilation | 28 days
Rate of ICU admission | 28 days
Rate and time of CRP,ES,Biochemical criterion(CK,ALT,Mb)recovery | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Institute of Infectious Disease, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided